CLINICAL TRIAL: NCT03095846
Title: Cold Induced Activation of Brown Fat in Winter Swimmers
Brief Title: Cold Induced Activation of Brown Adipose Tissue in Winter Swimmers
Acronym: COLDBAT_WS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanna Søberg, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: H-16038581-COLDBAT_WS
Record Dates: First submitted 2017-03-06; First posted 2017-03-30 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Adipose Tissue; Brown Adipose Tissue; Brown Fat; Uncoupling Protein 1; Adipokines; Proteomics; Infra-red Thermography; BAT; Winter Swimmers; Type2 Diabetes; Proteins
MeSH Terms: interventions — Cool-Down Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Winter Swimmers (Experimental): Individualized cooling protocol
  Interventions: Procedure: Cooling
- Not-winter Swimmers (Experimental): Individualized cooling protocol
  Interventions: Procedure: Cooling

INTERVENTIONS:
Procedure: Cooling — Individualized cooling protocol
  Other Names: Cold activation; Cold stimulation; Cold activation of BAT

SUMMARY:
This study investigates cold-induced brown fat activation in winter swimmers and not-winter swimmers by skin temperature measures assessed with infra red thermography imaging and skin temperatures. Winter swimmers and not-winter swimmers will participate in an acute cooling intervention and thermoneutral intervention for comparison of energy expenditure and skin temperatures at the supraclavicular area.

DETAILED DESCRIPTION:
The field of human brown adipose tissue (BAT) research is focused on activation of BAT as a means of manipulating energy expenditure and potentially anti-obesity and anti-diabetic properties of the tissue. This is well established in rodent studies and explained as due to the specific brown fat uncoupling protein 1 (UCP1). Despite increasing evidence that indicates a metabolic regulatory role of BAT in humans, BAT activation/recruitment is not fully understood.

Cold induced brown fat activity will be measured by skin temperature measures by means of infra-red thermography imaging and skin temperature.

15 healthy male winter swimmers and 8 healthy male non-winter swimmers (controls) will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

Age 18-35 years. Men Caucasian white Body Mass Index 19-25 kg/m2. Moderate physical activity level (not more than 8-10 hours of training pr. Week) Ability to give informed consent. Ability to follow verbal and written instructions in Danish. Body fat percent under 21% measured at the pre-examination day. Winter swimmers: Min. 2 swim/ week. Swimming in winter-season in open water outdoor in Denmark from September/October until study start in March.

Not-winter swimmers: Not winter-swimmers or taken cold showers on a regular basis.

Exclusion Criteria:

* Chronic diseases: Hormonal: Metabolic Diseases mb. Graves, hypothyroidism, myxedema and goiter. Diabetes Melitus, Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure), cancer treated within last 3 years.

Tobacco, marijuana or intravenous drug use within 1 year of screening. Dieting, recent weight loss (>3 kg within 3 month) or a history of an eating disorder.

Dietary supplements. History of depression, psychosis, or other psychiatric illness requiring hospitalization.

Alcohol consumption >14 units/week. History of alcohol abuse within the past 3 years. Known liver disease or elevated liver biomarkers more than 2 times upper normal levels in the preliminary investigation.

Known kidney disease or elevated kidney biomarkers, in the preliminary investigation.

Use of daily medications, except for seasonal use of antihistamines. Diagnosed sleep disturbances.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
5. Difference in brown adipose tissue (BAT) activity after cooling between Winter Swimmers (WS) and No-Winter Swimmers (NWS). | Difference in peak temperature after 2 hours of cooling.
  BAT activity is measured by skin temperature in the supraclavicular BAT depot using infrared thermography imaging. Difference between peak temperature change (peak temperature minus baseline temperature) during 2 hours of cooling is calculated.

SECONDARY OUTCOMES:
Difference in glucose control between WS and NWS. | Difference in glucose control between WS and NWS after a 2 hours glucose tolerance test under thermoneutral conditions.
  Difference in glucose control between WS and NWS in an oral glucose tolerance test measured as incremental area under the curve (iAUC).
Difference in resting energy expenditure after cooling versus no cooling | Difference in resting energy expenditure after 2 hours of cooling versus 2 hours of no cooling.
  Difference in resting energy expenditure after cooling versus no cooling between WS and NWS measured as mean difference in kilojoule per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Søberg, MSc., Principal Investigator — Center for Inflammation and Metabolism/Center for Physical Activity Research
Locations (1):
- Center for Inflammation and Metabolism/ Center for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No